CLINICAL TRIAL: NCT04877028
Title: Frailty Screening in the Swedish Emergency Department Setting
Status: Completed | Type: Observational
Sponsor: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Daniel Wilhelms, Principal Investigator, University Hospital, Linkoeping
Other Study IDs: 2021-00875FSSED
Record Dates: First submitted 2021-05-01; First posted 2021-05-07 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Frailty; Frailty Syndrome; Emergency Department; Geriatric Assessment; CFS
MeSH Terms: conditions — Frailty; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This prospective observational study will investigate the correlation of frailty in relation to serious outcomes. Serious outcomes are defined as: mortality within 30 days, admission to hospital, length of stay in the Emergency Department(ED), in hospital length of stay and revisits to the ED.

The exposure, frailty, will be assessed according to Clinical Frailty Scale. ED patients >65 years of age in a Swedish regional health care system (Region Östergötland, Sweden) comprising three EDs in Linköping, Norrköping and Motala. The outcomes will be compared according to the degree of frailty and censored over 7, 30 and 90 days respectively.

DETAILED DESCRIPTION:
Frailty is a common clinical syndrome in older adults that carries an increased risk for poor health outcomes including falls, incident disability, hospitalization, and mortality.

The clinical frailty scale (CFS) is a measure of frailty based on clinical judgement in a 9 level scale, categorized as "vulnerable" (1-4), "mildly frail" (5), moderatly frail (6) and severely and very severely frail (7-8).". A validation study of the CFS in community-dwelling older people showed that it performed better than measures of cognition, function or comorbidity in assessing risk for death. In a prospective observational study including consecutive ED patients aged 65 years or older The Hosmer-Lemeshow test indicated a good agreement between predicted probability and observed frequency of 30-day mortality and ICU admission.

The aim of this study will be to investigate if the fraily, assessed according to CFS, is associated with increased 30-day mortality. in a Swedish Emergency Care context. Secondary outcomes included 7-and 90-day mortality, ED length of stay, hospital admission, hospital length of stay, subsequent falls and medication changes. Additionally, we collect data on morbidity and comorbidities to assess the association with the level of frailty. Since this is a multicenter study, possible geographic differences will be studied as well. Based on the results of this study, possible interventions could be identified to improve the care of the frail geriatric patients presenting at the ED.

ELIGIBILITY:
Inclusion Criteria:

* ≥65 years, able to answer any questions, alternatively have a proxy

Exclusion Criteria:

- Patients: <65 years

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients of all genders at the age of ≥65 years seeking medical care at the three ED instances in Region Östergötland.
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2021-11-14 (Actual); Study Completion 2021-11-14 (Actual)

PRIMARY OUTCOMES:
Mortality in 30 days | All cause mortality up to 90 days from index visit
  Investigate level of mortality in cohort at 30 days

SECONDARY OUTCOMES:
Mortality in 7 and 90 days | All cause mortality up to 90 days from index visit
  Investigate level of mortality in cohort at 7 and 90 days
Admission to hospital | Hospital admission on index visit, censored at 90 days
  Investigate level of all cause admissions in cohort
ED length of stay | Length of stay at ED, censored at 4 days
  Investigate length of stay at ED
Hospital length of stay | Hospital length of stay from index visit, censored at 90 days
  Investigate hospital length of stay
Revisitis to the ED | Number of newly registered visits to the emergency department after index visit, censored at 90 days
  Number of newly registered visits to the emergency department after index visit
Fall prevalence after the index visit | Falls that resulted in further ED visits after index visit, censored in 90 days
  Falls that resulted in further ED visits
Alterations in medication during the visit (based on codes for Anatomical, Therapeutic, Chemical classification (ATC-code)) | Alterations in medications from index visit and during the follow-up period, censored at 90 days
  Alterations in medication and during the follow-up period

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Linköping, Linköping, Östergötland County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rockwood K, Song X, MacKnight C, Bergman H, Hogan DB, McDowell I, Mitnitski A. A global clinical measure of fitness and frailty in elderly people. CMAJ. 2005 Aug 30;173(5):489-95. doi: 10.1503/cmaj.050051. PMID 16129869
- [Background] Xue QL. The frailty syndrome: definition and natural history. Clin Geriatr Med. 2011 Feb;27(1):1-15. doi: 10.1016/j.cger.2010.08.009. PMID 21093718
- [Background] Rockwood K, Theou O. Using the Clinical Frailty Scale in Allocating Scarce Health Care Resources. Can Geriatr J. 2020 Sep 1;23(3):210-215. doi: 10.5770/cgj.23.463. eCollection 2020 Sep. PMID 32904824
- [Background] Wallis SJ, Wall J, Biram RW, Romero-Ortuno R. Association of the clinical frailty scale with hospital outcomes. QJM. 2015 Dec;108(12):943-9. doi: 10.1093/qjmed/hcv066. Epub 2015 Mar 15. PMID 25778109
- [Background] Kaeppeli T, Rueegg M, Dreher-Hummel T, Brabrand M, Kabell-Nissen S, Carpenter CR, Bingisser R, Nickel CH. Validation of the Clinical Frailty Scale for Prediction of Thirty-Day Mortality in the Emergency Department. Ann Emerg Med. 2020 Sep;76(3):291-300. doi: 10.1016/j.annemergmed.2020.03.028. Epub 2020 Apr 24. PMID 32336486
- [Derived] Munir Ehrlington S, Horlin E, Toll John R, Wretborn J, Wilhelms D. Frailty is associated with 30-day mortality: a multicentre study of Swedish emergency departments. Emerg Med J. 2024 Aug 21;41(9):514-519. doi: 10.1136/emermed-2023-213444. PMID 39053972